CLINICAL TRIAL: NCT04951622
Title: Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Nipocalimab Administered to Adults With Generalized Myasthenia Gravis
Brief Title: A Study of Nipocalimab Administered to Adults With Generalized Myasthenia Gravis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR109046; MOM-M281-011 (Other: Janssen Research & Development, LLC); 2020-005732-29 (EudraCT Number); 2023-504152-97-00 (Registry Identifier: EUCT number)
Expanded Access: NCT05221619 (Temporarily not available)
Record Dates: First submitted 2021-06-30; First posted 2021-07-07 (Actual); Results first posted 2025-07-23 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Nipocalimab (Experimental): Double-blind Placebo-controlled Phase: Participants will receive nipocalimab intravenous (IV) infusions once every 2 weeks (q2w) up to 24 weeks during double-blind placebo-controlled phase.
  Open-label Extension (OLE) Phase: Participants who complete the double-blind placebo-controlled phase will enter the OLE phase and continue to receive nipocalimab q2w IV infusion till study end.
  Interventions: Drug: Nipocalimab
- Placebo (Placebo Comparator): Double-blind Placebo-controlled Phase: Participants will receive matching placebo of nipocalimab IV infusion q2w up to 24 weeks during double-blind placebo-controlled phase.
  Interventions: Drug: Placebo
- Nipocalimab Subcutaneous (SC) (Experimental): OLE Phase: Participants from Cohort 1 will receive nipocalimab subcutaneous liquid in vial (SC-LIV) qw until Week 8. Participants with gMG from Cohort 2 who have not received nipocalimab previously, will receive nipocalimab SC-LIV until Week 8. Participants who complete the 8-week treatment period will have the opportunity to continue receiving nipocalimab SC-LIV qw in the Long term extension (LTE) period.
  Interventions: Drug: Nipocalimab SC-LIV

INTERVENTIONS:
Drug: Nipocalimab — Nipocalimab will be administered as an IV infusion.
  Other Names: JNJ-80202135, M281
  Arms: Nipocalimab
Drug: Placebo — Matching placebo will be administered as an IV infusion.
  Arms: Placebo
Drug: Nipocalimab SC-LIV — Nipocalimab will be administered subcutaneously.
  Arms: Nipocalimab Subcutaneous (SC)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of nipocalimab compared to placebo in participants with generalized myasthenia gravis (gMG). The purpose of the U.S. substudy is to evaluate how well it works in the body (pharmacodynamic [PD]) when given as an injection under the skin (subcutaneous) compared to when given through a vein (intravenous) in participants with gMG.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of myasthenia gravis (MG) with generalized muscle weakness meeting the clinical criteria for generalized myasthenia gravis (gMG) as defined by the Myasthenia Gravis Foundation of America (MGFA) Clinical Classification Class II a/b, III a/b, or IVa/b at screening
* Myasthenia Gravis - Activities of Daily Living (MG-ADL) score of greater than or equal to (>=) 6 at screening and baseline
* Has sufficient venous access to allow drug administration by infusion and blood sampling as per the protocol
* A woman of childbearing potential must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at screening and a negative urine pregnancy test at Day 1 prior to administration of study intervention
* A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum 90 days after receiving the last administration of study intervention
* For the SC Substudy (Cohort 1): Has reasonable abdominal skin area for SC administration
* For the SC Substudy (Cohort 1): Participants must be willing to comply with maintaining their stable dose of corticosteroids and/or immunosuppressants for the initial 8 weeks of the SC substudy, that is, through the SC Week 8 visit

Exclusion Criteria:

* Has any confirmed or suspected clinical immunodeficiency syndrome not related to treatment of his/her gMG, or has a family history of congenital or hereditary immunodeficiency unless confirmed absent in the participant
* Has MGFA Class I disease or presence of MG crisis (MGFA Class V) at screening, history of MG crisis within 1 month of screening, or fixed weakness (and/or 'burnt out' MG)
* Has had a thymectomy within 12 months prior to screening, or thymectomy is planned during the study
* Has known allergies, hypersensitivity, or intolerance to nipocalimab or its excipients
* Has experienced myocardial infarction, unstable ischemic heart disease, or stroke within 12 weeks of screening
* For the SC Substudy (Cohort 1): Participants who have undergone a recent tapering of their concomitant MG medication in the OLE
* For the SC Substudy (Cohort 1): Participants actively deteriorating at the SC Dose 1 visit for the SC substudy such that they meet the criteria for Clinical Deterioration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2026-04-17 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (111):
- United States (24):
  - Neuromuscular Research Center and Clinic, Paradise Valley, Arizona
  - HonorHealth Neurology, Scottsdale, Arizona
  - University of Southern California, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Care Access Research, Pasadena, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - FM Clinical Research, LLC South Florida Neurology Associates, P. A., Boca Raton, Florida
  - University of Florida Health Jacksonville, Jacksonville, Florida
  - Medsol Clinical Research Center Inc, Port Charlotte, Florida
  - University of South Florida, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - St. Elizabeth Medical Center, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Washington University School Of Medicine, St Louis, Missouri
  - Duke University School of Medicine, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Wesley Neurology, Cordova, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Vermont, Burlington, Vermont
- Australia (2):
  - Melbourne Neurology Group, North Melbourne
  - Gold Coast University Hospital, Southport
- Belgium (5):
  - ULB Hôpital Erasme, Anderlecht
  - AZ Sint Jan Brugge Oostende AV, Bruges
  - Cliniques Universitaires Saint Luc, Brussels
  - AZ Sint-Lucas, Ghent
  - University Hospitals Leuven, Leuven
- Canada (3):
  - The Ottawa Hospital Research Institute, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - McGill University, Montreal, Quebec
- China (14):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing
  - Xuanwu Hospital ,Capital Medical University, Beijing
  - Beijing Hospital, Beijing
  - The First Bethune Hospital of Jilin University, Changchun
  - Xiangya Hospital Central South University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Fujian Medical University Union Hospital, Fuzhou
  - The First Affiliated Hospital of Guangzhou University of Traditional Chinese Medicine, Guangzhou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - Qianfoshan hospital of Shandong Province, Jinan
  - Qilu Hospital of Shandong University, Jinan
  - Huashan Hospital Fudan University, Shanghai
  - Tianjin Medical University General Hospital, Tianjin
  - The Second Affiliated Hospital of Air Force Medical University - Tangdu Hospital, Xi'an
- Czechia (3):
  - Neurologie a rehabilitace Skopalíkova, Brno
  - Fakultni nemocnice Brno, Brno
  - Vseobecna Fakultní Nemocnice, Prague
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Rigshospitalet, København Ø
- France (4):
  - Hopital Pierre Wertheimer, Bron
  - CHU Grenoble, Grenoble
  - Hopital de la Pitie Salpetriere, Paris
  - Hopital PASTEUR, Provence-Alpes-Côte d'Azur
- Germany (6):
  - NeuroCure Clinical Research Center, Berlin
  - Universitatsmedizin Gottingen, Göttingen
  - Universitaetsklinikum Leipzig, Leipzig
  - Universitatsklinikum Schleswig Holstein Campus Lubeck, Lübeck
  - Universitatsklinikum Ulm, Ulm
  - DKD HELIOS Klinik Wiesbaden, Fachbereich Neurologie, Wiesbaden
- Italy (7):
  - U.O.P.I. di Psichiatria, Catania
  - Fondazione Istituto G. Giglio, Cefalù
  - Istituto Neurologico Carlo Besta, Milan
  - Azienda Ospedaliera Univ.- Università Degli studi della Campania - Luigi Vanvitelli, Napoli
  - IRCCS C. Mondino, Istituto Neurologico Nazionale, Fondazione, Pavia
  - Azienda ospedaliera Sant'Andrea di Roma- Università di Roma La Sapienza, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
- Japan (16):
  - Chiba University Hospital, Chiba
  - General Hanamaki Hospital, Hanamaki
  - Hiroshima University Hospital, Hiroshima
  - Teikyo University Hospital, Itabashi Ku
  - St Marianna University Hospital, Kawasaki Shi
  - Kagawa University Hospital, Kita Gun
  - Kumamoto University Hospital, Kumamoto
  - Iwate Medical University Hospital, Morioka
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - Niigata City General Hospital, Niigata
  - Hyogo College of Medicine Hospital, Nishinomiya-Shi
  - Sapporo Medical University Hospital, Sapporo
  - Hokkaido Medical Center, Sapporo
  - National Hospital Organization Sendai Medical Center, Sendai
  - Tokushima University Hospital, Tokushima
  - Tokyo Medical University Hospital, Tokyo
- Mexico (3):
  - iBiomed Research Unit, Aguascalientes
  - Consultorio Dr. Miguel Cortes, Cuernavaca
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara
- Poland (5):
  - Neurocentrum Bydgoszcz Sp Z O O, Bydgoszcz
  - NZOZ Wielospecjalistyczna Poradnia Lekarska 'Synapsis', Katowice
  - Centrum Neurologii Klinicznej Krakowska Akademia Neurologii, Krakow
  - Prywatny Gabinet Lekarski, Lublin
  - Centrum Medyczne NeuroProtect, Warsaw
- South Korea (4):
  - Pusan National University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Kyungpook National University Hospital, Daegu
  - Severance Hospital Yonsei University Health System, Seoul
- Spain (8):
  - Hosp. Gral. Univ. de Alicante, Alicante
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. de Basurto, Bilbao
  - Hosp. Virgen Macarena, Seville
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Univ. I Politecni La Fe, Valencia
- Sweden (2):
  - Karlstad Central Hospital, Karlstad
  - Karolinska Universitetssjukhuset Solna, Stockholm
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - Shin Kong Wu Ho Su Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency

REFERENCES:
- [Derived] Antozzi C, Fitzgibbon M. An evaluation of nipocalimab for the treatment of generalized myasthenia gravis. Expert Opin Biol Ther. 2025 Oct;25(10):1047-1058. doi: 10.1080/14712598.2025.2561935. Epub 2025 Sep 30. PMID 41021216
- [Derived] Raborn A, Savord A, Houts CR, Pease S, Scippa K, Ramchandren S. Psychometric analysis of the Neuro-QoL Fatigue in generalized Myasthenia Gravis (gMG) using data from a phase 3 trial. Qual Life Res. 2025 Sep;34(9):2577-2589. doi: 10.1007/s11136-025-03998-9. Epub 2025 Jun 14. PMID 40515798
- [Derived] Antozzi C, Vu T, Ramchandren S, Nowak RJ, Farmakidis C, Bril V, De Bleecker J, Yang H, Minks E, Park JS, Grudniak M, Smilowski M, Sevilla T, Hoffmann S, Sivakumar K, Suzuki Y, Youssef E, Sanga P, Karcher K, Zhu Y, Sheehan JJ, Sun H; Vivacity-MG3 Study Group. Safety and efficacy of nipocalimab in adults with generalised myasthenia gravis (Vivacity-MG3): a phase 3, randomised, double-blind, placebo-controlled study. Lancet Neurol. 2025 Feb;24(2):105-116. doi: 10.1016/S1474-4422(24)00498-8. PMID 39862879

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Results are currently reported for primary completion date (PCD, 17-Nov-2023). For open-label extension (OLE) phase, data for participants that were enrolled in OLE phase until the PCD is presented. OLE phase is still ongoing and complete results will be posted upon study completion.
Groups:
- Double Blind (DB) Phase: Placebo: During double blind (DB) phase, participants of present study received placebo matching to nipocalimab intravenous (IV) infusion as a loading dose on Day 1 (Week 0) followed by placebo matching to nipocalimab IV infusion as maintenance dose once every 2 weeks (q2w) from Week 2 up to Week 24.
- DB Phase: Nipocalimab: During DB phase, participants of present study received nipocalimab 30 milligrams per kilogram (mg/kg) IV infusion as a loading dose on Day 1 (Week 0) followed by nipocalimab 15 mg/kg IV infusion as maintenance dose once q2w from Week 2 up to Week 24.
- OLE Phase: Placebo to Nipocalimab: Present study participants who received placebo and completed DB phase entered OLE phase and received nipocalimab 15 mg/kg IV infusion q2w from OLE phase Day 1. Participants who discontinued DB treatment phase due to use of rescue medication for myasthenia gravis exacerbation or crisis were also eligible to enter the OLE phase.
- OLE Phase: Nipocalimab: Present study participants who received nipocalimab and completed DB phase entered OLE phase and received nipocalimab 15 mg/kg IV infusion q2w from OLE phase Day 1. Participants who discontinued DB treatment phase due to use of rescue medication for myasthenia gravis exacerbation or crisis were also eligible to enter the OLE phase.
- OLE Phase: Nipocalimab (MOM-M281-004 and MOM-M281-005): Participants who received nipocalimab in studies MOM-M281-004 (NCT03772587) and MOM-M281-005 (NCT03896295) entered OLE phase of the present study and received nipocalimab 15 mg/kg IV infusion q2w from OLE phase Day 1.
Period: DB Phase: Day 1 (Week 0) to Week 24
Arm/Group | Double Blind (DB) Phase: Placebo | DB Phase: Nipocalimab | OLE Phase: Placebo to Nipocalimab | OLE Phase: Nipocalimab | OLE Phase: Nipocalimab (MOM-M281-004 and MOM-M281-005)
Started | 99 | 100 | 0 | 0 | 0
Treated | 98 | 98 | 0 | 0 | 0
Completed | 82 | 87 | 0 | 0 | 0
Not Completed | 17 | 13 | 0 | 0 | 0
Not completed — Adverse Event | 7 | 5 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 2 | 0 | 0 | 0
Not completed — Death | 2 | 1 | 0 | 0 | 0
Not completed — Disease relapse | 0 | 1 | 0 | 0 | 0
Not completed — Progressive Disease | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0 | 0
Not completed — Randomized by mistake | 1 | 0 | 0 | 0 | 0
Not completed — Subject refused further study treatment | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0
Not completed — Failure to meet randomization criteria | 0 | 1 | 0 | 0 | 0
Period: OLE: Week 24 (OLE Day 1) up to 2 Years
Arm/Group | Double Blind (DB) Phase: Placebo | DB Phase: Nipocalimab | OLE Phase: Placebo to Nipocalimab | OLE Phase: Nipocalimab | OLE Phase: Nipocalimab (MOM-M281-004 and MOM-M281-005)
Started | 0 | 0 | 88 (Includes participants who discontinued DB phase due to use of rescue therapy.) | 88 (Includes participants who discontinued DB phase due to use of rescue therapy.) | 20
Treated | 0 | 0 | 88 | 88 | 19
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 88 | 88 | 20
Not completed — Adverse Event | 0 | 0 | 5 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 5 | 1
Not completed — Lack of Efficacy | 0 | 0 | 3 | 7 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 1 | 0
Not completed — Ongoing | 0 | 0 | 77 | 74 | 15
Not completed — Met eligibility criteria but discontinued during the screening period (not treated) | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomized participants who received at least 1 dose (partial or complete) of any study intervention in the double-blind phase. The safety analysis set (OL) included all participants who received at least 1 dose (partial or complete) of nipocalimab in the OLE phase
Groups:
- Total: Total of all reporting groups
Arm/Group | Double Blind (DB) Phase: Placebo | DB Phase: Nipocalimab | OLE Phase: Nipocalimab (MOM-M281-004 and MOM-M281-005) | Total
Number analyzed (Participants) | 98 | 98 | 19 | 215
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.7 (15.60) | 52.9 (15.49) | 52.7 (17.69) | 52.8 (15.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 66 | 10 | 132
  Male | 42 | 32 | 9 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 10 | 5 | 21
  Not Hispanic or Latino | 89 | 87 | 14 | 190
  Unknown or Not Reported | 3 | 1 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 29 | 28 | 0 | 57
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 65 | 66 | 19 | 150
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Double-blind (DB) Phase: Average Change From Baseline in Myasthenia Gravis - Activities of Daily Living (MG-ADL) Total Score Over Weeks 22, 23, and 24
Description: Average change from baseline over multiple timepoints (Weeks 22, 23, and 24) was reported in this outcome measure. The MG-ADL provided a rapid assessment of the participant's MG symptom severity of eight functions (talking, chewing, swallowing, breathing, impairment of ability to brush teeth or comb hair, impairment of ability to arise from a chair, double vision, eyelid droop) rated on a 4-point scale ranging from 0 (normal) to 3 (severe). MG-ADL total score was sum of 8 individual items, which ranging from 0 to 24. A higher score indicated greater symptom severity. Baseline was defined as the average of the screening and Day 1 total scores.
Time Frame: Baseline, Weeks 22, 23, and 24
Population: Primary efficacy analysis set included all randomized seropositive (with anti- acetylcholine receptor positive, anti muscle-specific kinase positive, and/or anti- lipoprotein-related protein receptor 4 positive) participants who received at least 1 dose (partial or complete) of any study intervention in the double-blind phase. Here, 'N' (overall number of participants analysed) signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Double Blind (DB) Phase: Placebo | DB Phase: Nipocalimab
Number analyzed (Participants) | 76 | 77
Score on a scale | -3.25 (0.335) | -4.70 (0.329)
Statistical Analysis 1: Comparison: Double Blind (DB) Phase: Placebo vs DB Phase: Nipocalimab; Test type: Superiority; p = 0.002, mixed effects model for repeated measure; Difference of LS Means = -1.45, 95% CI 2-sided [-2.38 to -0.52], Standard Error of Mean 0.47

2. Secondary Outcome: DB Phase: Average Change From Baseline in Quantitative Myasthenia Gravis (QMG) Score Over Weeks 22 and 24
Time Frame: Baseline, Weeks 22, and 24
Reporting Status: Not Posted, anticipated posting 2027-04

3. Secondary Outcome: DB Phase: Percentage of Participants Who Had Achieved at Least a 2-point Average Improvement From Baseline in Myasthenia Gravis - Activities of Daily Living (MG-ADL) Total Score Over Weeks 22, 23, and 24
Time Frame: Weeks 22, 23, and 24
Reporting Status: Not Posted, anticipated posting 2027-04

4. Secondary Outcome: DB Phase: Percentage of Participants Who Had Achieved an Improvement of Greater Than or Equal to (>=) 2 Points in the Myasthenia Gravis - Activities of Daily Living (MG-ADL) Total Score at Week 1 and/or Week 2
Time Frame: Weeks 1 and 2
Reporting Status: Not Posted, anticipated posting 2027-04

5. Secondary Outcome: DB Phase: Percentage of Participants Who Had an Improvement of >= 2 Points in the MG-ADL Total Score From Week 4 Through Week 24 With no More Than 2 Non-consecutive Excursions Allowed Between Weeks 6 Through 23
Time Frame: From Week 4 up to Week 24
Reporting Status: Not Posted, anticipated posting 2027-04

6. Secondary Outcome: DB Phase: Percentage of Participants Who Had Achieved at Least a 50 Percent (%) Average Improvement From Baseline in the Myasthenia Gravis - Activities of Daily Living (MG-ADL) Total Score Over Weeks 22, 23, and 24
Time Frame: Weeks 22, 23, and 24
Reporting Status: Not Posted, anticipated posting 2027-04

7. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Time Frame: From start of treatment (DB phase Day 1) up to 4 years 9 months
Reporting Status: Not Posted, anticipated posting 2027-04

8. Secondary Outcome: Percentage of Participants With Treatment-emergent Serious Adverse Events (TESAEs)
Time Frame: From start of treatment (DB phase Day 1) up to 4 years 9 months
Reporting Status: Not Posted, anticipated posting 2027-04

9. Secondary Outcome: Percentage of Participants With AEs of Special Interest (AESIs)
Time Frame: From start of treatment (DB phase Day 1) up to 4 years 9 months
Reporting Status: Not Posted, anticipated posting 2027-04

10. Secondary Outcome: Number of Participants With Change in Vital Signs
Time Frame: From start of treatment (DB phase Day 1) up to 4 years 9 months
Reporting Status: Not Posted, anticipated posting 2027-04

11. Secondary Outcome: Number of Participants With Change in Clinical Laboratory Values
Time Frame: From start of treatment (DB phase Day 1) up to 4 years 9 months
Reporting Status: Not Posted, anticipated posting 2027-04

12. Secondary Outcome: Number of Participants With Change From Baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) Score
Time Frame: From start of treatment (Day 1) up to 4 years 9 months
Reporting Status: Not Posted, anticipated posting 2027-04

13. Secondary Outcome: DB Phase: Percentage of Participants Who Had an Improvement of >= 3 Points in Quantitative Myasthenia Gravis (QMG) Score From Baseline, at Week 2 Through Week 24, With No More Than 2 Non-consecutive Excursions Allowed Between at Weeks 4 Through Week 22
Time Frame: Baseline, Week 2 up to Week 24
Reporting Status: Not Posted, anticipated posting 2027-04

14. Secondary Outcome: DB Phase: Average Change From Baseline in the Fatigue Items of the Quality of Life in Neurological Disorders (Neuro-QoL) Fatigue Scale Total Score Over Weeks 22 and 24
Time Frame: Baseline up to Weeks 22, and 24
Reporting Status: Not Posted, anticipated posting 2027-04

15. Secondary Outcome: DB Phase: Average Change From Baseline in the Revised Myasthenia Gravis Quality of Life (Revised) Instrument (MG-Qol15r) Score Over Weeks 22 And 24
Time Frame: Baseline up to Weeks 22, and 24
Reporting Status: Not Posted, anticipated posting 2027-04

16. Secondary Outcome: DB Phase: Change From Baseline in the Visual Analog Scale (VAS) Score of European Quality of Life (EuroQol) 5-Dimension 5-Level (EQ-5D-5L) Scale Over 24 Weeks
Time Frame: Baseline up to Week 24
Reporting Status: Not Posted, anticipated posting 2027-04

17. Secondary Outcome: DB Phase: Change From Baseline in the Health Status Index of the EuroQol 5-Dimension 5-Level (EQ-5D-5L) Scale Over 24 Weeks
Time Frame: Baseline up to Week 24
Reporting Status: Not Posted, anticipated posting 2027-04

18. Secondary Outcome: DB Phase: Percentage of Participants With Myasthenia Gravis - Activities of Daily Living (MG-ADL) Score of 0 or 1 Over Time
Time Frame: Baseline up to Week 24
Reporting Status: Not Posted, anticipated posting 2027-04

19. Secondary Outcome: DB Phase: Percentage of Participants With Myasthenia Gravis - Activities of Daily Living (MG-ADL) Score of 0 or 1 at Any Time
Time Frame: Baseline up to Week 24
Reporting Status: Not Posted, anticipated posting 2027-04

20. Secondary Outcome: DB Phase: Percentage of Participants With Myasthenia Gravis - Activities of Daily Living (MG-ADL) Score of 0 or 1 at 50% of Timepoints
Time Frame: Baseline up to Week 24
Reporting Status: Not Posted, anticipated posting 2027-04

21. Secondary Outcome: DB Phase: Percentage of Participants With Myasthenia Gravis - Activities of Daily Living (MG-ADL) Score of 0 or 1 at 75% of Timepoints
Time Frame: Baseline up to Week 24
Reporting Status: Not Posted, anticipated posting 2027-04

22. Secondary Outcome: Serum Concentrations of Nipocalimab Over Time
Time Frame: DB Phase: Predose and 45 minutes post-dose on Day 1, Weeks 2, 4, 8, 12,16, 20, 24;OL Phase: Predose on Day 1, Weeks 8, 16, 24, 36, 48, 60, 72, 84, and 96
Reporting Status: Not Posted, anticipated posting 2027-04

23. Secondary Outcome: Number of Participants With Antibodies to Nipocalimab (Anti-Drug Antibodies [ADAs] and Neutralizing Antibodies [NAbs])
Time Frame: From start of treatment (Day 1) up to 4 years 9 months
Reporting Status: Not Posted, anticipated posting 2027-04

24. Secondary Outcome: Percent Change From Baseline in Total Serum Immunoglobulin G (IgG) Concentrations
Time Frame: Baseline up to 4 years 9 months
Reporting Status: Not Posted, anticipated posting 2027-04

25. Secondary Outcome: Change From Baseline in Levels of Autoantibodies Associated With Generalized Myasthenia Gravis (gMG)
Time Frame: Baseline up to 4 years 9 months
Reporting Status: Not Posted, anticipated posting 2027-04

26. Secondary Outcome: Change From Baseline in Myasthenia Gravis - Activities of Daily Living (MG-ADL) Score as a Function of IgG
Time Frame: Baseline up to 4 years 9 months
Reporting Status: Not Posted, anticipated posting 2027-04

27. Secondary Outcome: Change From Baseline in Quantitative Myasthenia Gravis (QMG) Score as a Function of Immunoglobulin G (IgG)
Time Frame: Baseline up to 4 years 9 months
Reporting Status: Not Posted, anticipated posting 2027-04

28. Secondary Outcome: Change From Baseline in Myasthenia Gravis - Activities of Daily Living (MG-ADL) Score as a Response to Percent Change in Autoantibody Levels in Seropositive Participants Treated With Nipocalimab
Time Frame: Baseline up to 4 years 9 months
Reporting Status: Not Posted, anticipated posting 2027-04

29. Secondary Outcome: Change From Baseline in QMG Score as a Response to Percent Change in Autoantibody Levels in Seropositive Participants Treated With Nipocalimab
Time Frame: Baseline up to 4 years 9 months
Reporting Status: Not Posted, anticipated posting 2027-04

ADVERSE EVENTS:
Time Frame: DB: All-cause mortality: From screening (Day -28) to Week 24; SAE and other AEs: From Day 1 (Week 0) to Week 24; OLE: From Week 24 (OLE Day 1) up to 2 years
Description: DB: SAE and Other AEs: Safety analysis set included all participants who received at least 1 dose (partial or complete) of any study intervention in the DB phase. All cause-mortality: Randomized analysis set included all participants who were randomized in the study. OLE: The safety analysis set included all participants who received at least 1 dose (partial or complete) of nipocalimab in the OLE phase. OLE phase analysis is until PCD and final results will be posted upon study completion.
Groups:
- OLE Phase: Nipocalimab (MOMM281- 004 and MOM-M281-005): Participants who received nipocalimab in studies MOM-M281-004 (NCT03772587) and MOM-M281-005 (NCT03896295) entered OLE phase of the present study and received nipocalimab 15 mg/kg IV infusion q2w from OLE phase Day 1.
Arm/Group | Double Blind (DB) Phase: Placebo | DB Phase: Nipocalimab | OLE Phase: Placebo to Nipocalimab | OLE Phase: Nipocalimab | OLE Phase: Nipocalimab (MOMM281- 004 and MOM-M281-005)
All-Cause Mortality (participants affected / at risk) | 2/99 | 1/100 | 1/88 | 1/88 | 1/19
Serious Adverse Events (participants affected / at risk) | 14/98 | 9/98 | 10/88 | 16/88 | 7/19
Other Adverse Events (participants affected / at risk) | 65/98 | 69/98 | 57/88 | 59/88 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind (DB) Phase: Placebo (N=98) | DB Phase: Nipocalimab (N=98) | OLE Phase: Placebo to Nipocalimab (N=88) | OLE Phase: Nipocalimab (N=88) | OLE Phase: Nipocalimab (MOMM281- 004 and MOM-M281-005) (N=19)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Atrioventricular Block Complete (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiogenic Shock (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Hypertensive Heart Disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Myocardial Ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Grey Matter Heterotopia (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
Eyelid Pain (Eye disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Liver Disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Anaphylactic Shock (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Haemophagocytic Lymphohistiocytosis (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Coronavirus Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Escherichia Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis Salmonella (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes Zoster Oticus (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Perinephric Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 1 | 1 | 0
Pneumonia Aspiration (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia Bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Parathyroid Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Intracranial Mass (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Myasthenia Gravis (Nervous system disorders) | 4 | 3 | 1 | 6 | 2
Myasthenia Gravis Crisis (Nervous system disorders) | 2 | 1 | 1 | 0 | 1
Non-Epileptic Paroxysmal Event (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Toxic Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Major Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Nephropathy (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal Tubular Necrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind (DB) Phase: Placebo (N=98) | DB Phase: Nipocalimab (N=98) | OLE Phase: Placebo to Nipocalimab (N=88) | OLE Phase: Nipocalimab (N=88) | OLE Phase: Nipocalimab (MOMM281- 004 and MOM-M281-005) (N=19)
Anaemia (Blood and lymphatic system disorders) | 3 | 4 | 3 | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
White Blood Cell Disorder (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 1 | 1 | 1
Bundle Branch Block Left (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 2 | 1 | 0 | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Thyroid Mass (Endocrine disorders) | 0 | 0 | 0 | 1 | 2
Angle Closure Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eye Pain (Eye disorders) | 1 | 0 | 0 | 0 | 1
Eyelid Ptosis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 7 | 5 | 2 | 3
Diverticulum Intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Food Poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 5 | 4 | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 1
Asthenia (General disorders) | 2 | 0 | 1 | 0 | 1
Catheter Site Erythema (General disorders) | 0 | 0 | 0 | 0 | 1
Cyst (General disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 3 | 4 | 5 | 3 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 1 | 1
Infusion Site Bruising (General disorders) | 0 | 1 | 0 | 0 | 1
Infusion Site Erythema (General disorders) | 0 | 0 | 0 | 0 | 1
Infusion Site Extravasation (General disorders) | 1 | 0 | 0 | 0 | 1
Malaise (General disorders) | 1 | 1 | 0 | 0 | 1
Oedema (General disorders) | 1 | 0 | 1 | 0 | 1
Oedema Peripheral (General disorders) | 0 | 10 | 4 | 1 | 2
Pain (General disorders) | 0 | 1 | 0 | 0 | 1
Peripheral Swelling (General disorders) | 1 | 1 | 3 | 1 | 2
Pyrexia (General disorders) | 1 | 7 | 1 | 5 | 1
Secretion Discharge (General disorders) | 0 | 0 | 0 | 0 | 1
Swelling (General disorders) | 1 | 0 | 0 | 0 | 1
Swelling Face (General disorders) | 1 | 0 | 0 | 0 | 1
Hepatic Cyst (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 1
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Seasonal Allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 2 | 2 | 2 | 3
Covid-19 (Infections and infestations) | 9 | 11 | 7 | 7 | 5
Covid-19 Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastric Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 0 | 1
Gastrointestinal Viral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Helicobacter Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Herpes Ophthalmic (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 10 | 9 | 11 | 10 | 2
Oral Herpes (Infections and infestations) | 2 | 1 | 0 | 2 | 2
Pharyngitis (Infections and infestations) | 0 | 2 | 3 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 2 | 5 | 3 | 2
Tooth Infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 8 | 6 | 9 | 9 | 5
Urinary Tract Infection (Infections and infestations) | 0 | 5 | 9 | 8 | 2
Viral Diarrhoea (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Viral Infection (Infections and infestations) | 0 | 0 | 1 | 2 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 2 | 1
Animal Bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 3 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 2 | 3
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Muscle Hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Muscle Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Skin Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Blood Cholesterol Increased (Investigations) | 1 | 0 | 0 | 1 | 1
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 2 | 0 | 1 | 1
Blood Pressure Increased (Investigations) | 0 | 3 | 1 | 0 | 1
C-Reactive Protein Increased (Investigations) | 0 | 0 | 1 | 2 | 1
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 0 | 0 | 2 | 1
Haemoglobin Decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Intraocular Pressure Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Low Density Lipoprotein Increased (Investigations) | 1 | 0 | 1 | 3 | 1
Lymphocyte Count Decreased (Investigations) | 1 | 0 | 1 | 0 | 1
Monocyte Count Decreased (Investigations) | 1 | 0 | 1 | 0 | 1
Neutrophil Count Increased (Investigations) | 1 | 2 | 0 | 1 | 1
Sars-Cov-2 Test Positive (Investigations) | 0 | 1 | 2 | 1 | 2
Weight Increased (Investigations) | 0 | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2 | 4 | 4 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 8 | 4 | 9 | 1
Medial Tibial Stress Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 | 12 | 3 | 6 | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 | 5 | 2 | 4 | 4
Spinal Deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Diabetic Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 5 | 1 | 2 | 1
Dizziness Postural (Nervous system disorders) | 1 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 17 | 14 | 10 | 5 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 0 | 0 | 1
Loss of Consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Lumbar Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 1 | 0 | 1 | 1
Myasthenia Gravis (Nervous system disorders) | 9 | 9 | 5 | 8 | 4
Paraesthesia (Nervous system disorders) | 0 | 2 | 1 | 0 | 1
Tremor (Nervous system disorders) | 1 | 2 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2 | 2
Insomnia (Psychiatric disorders) | 2 | 5 | 1 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Major Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Breast Haematoma (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 1 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Perioral Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 2 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 2 | 4 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2024-08-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT04951622/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT04951622/SAP_001.pdf